CLINICAL TRIAL: NCT01355679
Title: A Feasibility Trial Using Molecular-Guided Therapy for the Treatment of Patients With Refractory or Recurrent Neuroblastoma
Brief Title: Molecular Guided Therapy for Refractory or Recurrent Neuroblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giselle Sholler (Other)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Study Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NMTRC 001; NCT01375517 (obsolete NCT alias)
Record Dates: First submitted 2011-05-13; First posted 2011-05-18 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Guided therapy (Experimental): A total of 14 eligible neuroblastoma patients who are refractory or relapsed on conventional therapy will be treated. Guided therapy will allow the use of any therapeutic combination (up to 4 agents) provided it includes medications contained in the study report. All patients will be followed for survival, disease response, progression and safety. All patients will be treated according to the discretion of the treating oncologist and study committee (minimum 3 oncologists and one pharmacist). Extent of disease will be measured and assessed for changes throughout the course of the study and at 6-8 week intervals (every 2 cycles).
  Interventions: Device: Guided Therapy

INTERVENTIONS:
Device: Guided Therapy — A total of 14 eligible neuroblastoma patients who are refractory or relapsed on conventional therapy will be treated. Guided therapy will allow the use of any therapeutic combination (up to 4 agents) provided it includes medications contained in the study report. All patients will be followed for disease response, progression and safety. All patients will be treated according to the discretion of the treating oncologist and study committee (minimum 3 oncologists and one pharmacist). Extent of disease will be measured and assessed for changes throughout the course of the study and at 6-8 week intervals (every 2 cycles).

SUMMARY:
The purpose of this study is to test the feasibility (ability to be done) of an experimental test to help plan your cancer treatment. This study plan is not studying the effectiveness of the proposed combinations of therapy for your cancer that you may receive after the experimental testing.

This study will look at an experimental technology to determine a tumor's molecular makeup (gene expression profile). This technology (called "OncInsights") is being used to discover new ways to understand cancers and potentially predict the best treatments for patients with cancer in the future. The experimental technology has not been approved by the U.S. Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven neuroblastoma and confirmation of refractory or recurrent disease with histologic confirmation at diagnosis or at the time of recurrence/progression
* Patients must be age > 12 months and ≤ 21 at initial diagnosis.
* Life expectancy must be more than 3 months
* If measurable disease, this must be demonstrated by residual abnormal tissue at a primary or metastatic site measuring more than 1 cm in any dimension by standardized imaging (CT or MRI); tumor must be accessible for biopsy. Patients with bone marrow only disease expected to be > 75% are eligible to enroll.
* Current disease state must be one for which there is currently no known curative therapy
* Lansky or KarnofskyScore must be more than 50
* Patients without bone marrow metastases must have an ANC > 750/μl and platelet count > 50,000/μl
* Adequate liver function must be demonstrated, defined as:

  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age AND
  * SGPT (ALT) < 10 x upper limit of normal (ULN) for age
* No other significant organ toxicity defined as > Grade 2 by National Cancer Institute Common Toxicity Criteria for Adverse Events NCI-CTCAE V4.0
* A negative serum pregnancy test is required for female participants of child bearing potential (≥ 13 years of age or after onset of menses)
* Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.
* Informed Consent: All patients and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines. Voluntary consent for optional biology studies will be included.

Exclusion Criteria:

* Patients who have received any chemotherapy within the last 7 days prior to enrollment and 14 days prior to study treatment start date.
* Patients who have received any radiotherapy within the last 30 days must have another site of disease to follow.
* Patients receiving anti-tumor therapy for their disease or any investigational drug concurrently
* Patients with serious infection or a life-threatening illness (unrelated to tumor) that is > Grade 2 (NCI CTCAE V4.0), or active, serious infections requiring parenteral antibiotic therapy.
* Patients with any other medical condition, including malabsorption syndromes, mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the interpretation of the results or which would interfere with a patient's ability to sign or the legal guardian's ability to sign the informed consent, and patient's ability to cooperate and participate in the study

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2013-09 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer at Atrium Health
Locations (7):
- United States (7):
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Arnold Palmer Hospital for Children- MD Anderson, Orlando, Florida
  - National Cancer Institute, Bethesda, Maryland
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina

REFERENCES:
- See also: Beat Childhood Cancer — https://beatcc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, multi-center prospective feasibility study in patients with refractory or recurrent neuroblastoma that enrolled at NMTRC centers across the country between 8/11/2011 and 11/26/2012.
Groups:
- Guided Therapy: A total of 14 neuroblastoma patients who are refractory or relapsed on conventional therapy will be treated. Guided therapy will allow the use of any therapeutic combination (up to 4 agents) provided it includes medications contained in the study report. All patients will be followed for survival, disease response, progression and safety. All patients will be treated according to the discretion of the treating oncologist and study committee (minimum 3 oncologists and one pharmacist). Extent of disease will be measured and assessed for changes throughout the course of the study and at 6-8 week intervals (every 2 cycles).
  Guided Therapy: A total of 14 neuroblastoma patients who are refractory or relapsed on conventional therapy will be treated. Guided therapy will allow the use of any therapeutic combination (up to 4 agents) provided it includes medications contained in the study report. All patients will be followed for disease response, progression and safety. All patients will be
Period: Overall Study
Arm/Group | Guided Therapy
Started | 16
Completed | 14
Not Completed | 2
Not completed — benign tumor types found at biopsy | 2

BASELINE CHARACTERISTICS:
Population: Multiply relapsed or refractory neuroblastoma.
Groups:
- Guided Therapy: All subjects receive guided therapy in therapeutic combination (up to 4 agents) provided it includes medications contained in the study report.
Arm/Group | Guided Therapy
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Are Able to Meet Feasibility Parameters.
Description: Feasibility parameter defined as: Enrollment onto study, quality mRNA obtained, gene chip completed, tumor board held, medical monitor review and approval, start of treatment by 21 days post biopsy/surgical resection date, and then completion of 1 cycle of therapy."
Time Frame: 1 year
Population: All subjects had soft tissue disease in which biopsy was possible. Two subjects were deemed ineligible due to benign tumor type after biopsy.
Measure: Number; unit: percentage of participants
Arm/Group | Guided Therapy
Number analyzed (Participants) | 14
percentage of participants | 100

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: To determine the safety of allowing a molecular tumor board to determine individualized treatment plans
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Guided Therapy
Number analyzed (Participants) | 14
participants | 12

3. Secondary Outcome: Overall Response Rate (ORR) of Participants Using RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Measure: Number; unit: percentage of participants with PR or CR
Arm/Group | Guided Therapy
Number analyzed (Participants) | 14
percentage of participants with PR or CR | 7

4. Secondary Outcome: Activity of Treatments Chosen Based on Progression Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Guided Therapy
Number analyzed (Participants) | 14
Days | 59 [43 to 59]

ADVERSE EVENTS:
Time Frame: Time on therapy plus 30 days after last dose and until all related events resolved, an average of 1 year.
Arm/Group | Guided Therapy
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 12/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guided Therapy (N=14)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
ALT elevation (Hepatobiliary disorders) | 2 (2)
AST Elevation (Hepatobiliary disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Elevated Bilirubin (Hepatobiliary disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Hypoalbunemia (Blood and lymphatic system disorders) | 2 (2)
Hypocalcemia (General disorders) | 1 (1)
Hypophosphatemia (General disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 7 (7)
Lymphocytopenia (Blood and lymphatic system disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 2 (2)
Myalgia (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 7 (7)
Pain (General disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight Loss (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No